CLINICAL TRIAL: NCT00194025
Title: Add-on Valproate in Late Life Schizophrenia
Brief Title: Valproate in Late Life Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Martha Sajatovic MD, Case Western Reserve University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10850-01-L0348
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2011-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Anticonvulsants; Valproic Acid; Valproate
MeSH Terms: conditions — Schizophrenia | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- valproate (Experimental): All participants received open-label, add-on valproate.
  Interventions: Drug: Valproate

INTERVENTIONS:
Drug: Valproate — Enrolled individuals received adjunctive, open-label valproate semisodium, initially started as valproate semisodium delayed -release 250 mg at bedtime for two weeks, then changed to valproate semisodium extended- release 500 mg at bedtime. Medication was administered on an outpatient/ambulatory basis, and adjusted as tolerated to target serum levels of 50-100 µg/mL. In cases where sedation or other side effects occurred, dosage was reduced. Valproate semisodium was prescribed in a single dose at bedtime.
  Other Names: Depakote; Depakote ER

SUMMARY:
The purpose of this research study is to analyze the effectiveness and tolerability of a medication, valproate ( Depakote and Depakote ER), in individuals age 50 years and older who have schizophrenia.

DETAILED DESCRIPTION:
It is known that up to 30% of individuals with schizophrenia continue to have symptoms even when treated with current FDA-approved medications intended to treat their schizophrenia. Anticonvulsant medications such as valproate (Depakote and Depakote ER) are known to be effective for related conditions such as bipolar disorder (manic depressive illness), and are also used by some physicians in clinical settings in combination with antipsychotic medications to treat symptoms of schizophrenia. Currently Depakote and Depakote ER are approved by the FDA to treat bipolar disorder and to treat seizure disorder. This study will test to see if Depakote and Depakote ER may improve symptoms of schizophrenia as well when added to antipsychotic medications.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of schizophrenia as confirmed by the MINI
* Must be on antipsychotic medication
* Must be age 50 year or older
* Must be capable of providing written informed consent for study participation. In situations where individuals have guardians of person, guardian and subject must both provide written consent; and
* Must live in the Northeast Ohio area.

Exclusion Criteria:

* A primary psychiatric DSM Axis I diagnosis other than schizophrenia
* Actively abusing substances; or
* Medically unstable.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-11; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University School of Medicine
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

REFERENCES:
- [Result] Sajatovic M, Coconcea N, Ignacio RV, Blow FC, Hays RW, Cassidy KA, Meyer WJ. Adjunct extended-release valproate semisodium in late life schizophrenia. Int J Geriatr Psychiatry. 2008 Feb;23(2):142-7. doi: 10.1002/gps.1854. PMID 17582828

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at an academic psychiatry clinic in the mid-western United States. Data was collected from participants from February 2004 to November 2006. Participants were recruited in response to self-referrals from advertisements and by referrals from mental health practitioners.
Groups:
- Valproate: Enrolled individuals received adjunctive, openlabel valproate semisodium, initially started as valproate semisodium delayed-release 250 mg at bedtime for two weeks, then changed to valproate semisodium extended-release 500 mg at bedtime. Medication was administered on an outpatient/ambulatory basis, and adjusted as tolerated to target serum levels of 50- 100 mg/mL. In cases where sedation or other side effects occurred, dosage was reduced. Valproate semisodium was prescribed in a single dose at bedtime.
Period: Overall Study
Arm/Group | Valproate
Started | 20 (The intent-to-treat population received at least one dose of valproate semisodium.)
Completed | 15 (5 participants withdrew prematurely)
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — non-adherence with study medication | 4

BASELINE CHARACTERISTICS:
Arm/Group | Valproate
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Schizophrenia Psychopathology as Assessed by the Positive and Negative Symptom Scale (PANSS)
Description: The best and worst possible overall PANSS scores are 30 and 210 units on a scale, respectively.
Time Frame: Baseline to 12 weeks
Population: Last Observation Carried Forward (LOCF) was used as the imputation technique.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Valproate
Number analyzed (Participants) | 20
scores on a scale | -17.45 (14.87)
Statistical Analysis 1: Comparison: Valproate; The 1 sided t-test was applied to the scores at baseline vs. the scores at 12 weeks; Test type: Superiority or Other; p < 0.001, t-test, 1 sided

2. Secondary Outcome: Change in Cognitive Status as Measured by the Mini-mental State Examination (MMSE)
Description: The best and worst possible overall scores are 31 and 0 units on a scale, respectively.
Time Frame: Baseline to 12 weeks
Population: Last Observation Carried Forward (LOCF) was used as the imputation technique.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Valproate
Number analyzed (Participants) | 20
scores on a scale | 0.4 (3.218)
Statistical Analysis 1: Comparison: Valproate; The 1 sided t-test was applied to the scores at baseline vs. the scores at 12 weeks; Test type: Superiority or Other; p = 0.585, t-test, 1 sided

3. Secondary Outcome: Change in Overall Functioning as Measured by the Global Assessment Scale (GAS)
Description: The best and worst possible GAS scores are 100 and 1 units on a scale, respectively.
Time Frame: Baseline to 12 weeks
Population: Last Observation Carried Forward (LOCF) was used as the imputation technique.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Valproate
Number analyzed (Participants) | 20
scores on a scale | 16.35 (15.09)
Statistical Analysis 1: Comparison: Valproate; The 1 sided t-test was applied to the scores at baseline vs. the scores at 12 weeks; Test type: Superiority or Other; p < 0.001, t-test, 1 sided

4. Secondary Outcome: Change in Depression Symptoms as Measured by the Geriatric Depression Scale (GDS)
Description: The best and worst possible GDS scores are 0 and 30 units on a scale, respectively.
Time Frame: Baseline to 12 weeks
Population: Last Observation Carried Forward (LOCF) was used as the imputation technique.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Valproate
Number analyzed (Participants) | 18
scores on a scale | -1.556 (2.502)
Statistical Analysis 1: Comparison: Valproate; The 1 sided t-test was applied to the scores at baseline vs. the scores at 12 weeks; Test type: Superiority or Other; p = 0.017, t-test, 1 sided

5. Secondary Outcome: Change in Overall Mental Health Status as Measure by the Mental Composite Score (MCS) Subscale of the Short Form 36 Health Survey (SF-36)
Description: The best and worst possible MCS scores are 100 and 1 units on a scale, respectively.
Time Frame: Baseline to 12 weeks
Population: The number of participants for analysis was based on available data. Last Observation Carried Forward (LOCF) was used as the imputation technique.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Valproate
Number analyzed (Participants) | 14
scores on a scale | 5.298 (7.968)
Statistical Analysis 1: Comparison: Valproate; The 1 sided t-test was applied to the scores at baseline vs. the scores at 12 weeks; Test type: Superiority or Other; p = 0.027, t-test, 1 sided

6. Secondary Outcome: Change in Physical Health Status as Measure by the Physical Composite Score (PCS) Subscale of the Short Form 36 Health Survey (SF-36)
Description: The best and worst possible PCS scores are 100 and 0 units on a scale, respectively.
Time Frame: Baseline to 12 weeks
Population: Last Observation Carried Forward (LOCF) was used as the imputation technique.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Valproate
Number analyzed (Participants) | 14
scores on a scale | 0.932 (5.971)
Statistical Analysis 1: Comparison: Valproate; The 1 sided t-test was applied to the scores at baseline vs. the scores at 12 weeks; Test type: Superiority or Other; p = 0.569, t-test, 1 sided

7. Secondary Outcome: Change in Extrapyramidal Symptoms as Assessed by the Abnormal Involuntary Movement Scale (AIMS)
Description: The best and worst possible overall scores are 0 and 28 units on a scale, respectively.
Time Frame: Baseline to 12 weeks
Population: Last Observation Carried Forward (LOCF) was used as the imputation technique.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Valproate
Number analyzed (Participants) | 19
scores on a scale | -2.105 (4.108)
Statistical Analysis 1: Comparison: Valproate; The 1 sided t-test was applied to the scores at baseline vs. the scores at 12 weeks; Test type: Superiority or Other; p = 0.038, t-test, 1 sided

8. Secondary Outcome: Change in Extrapyramidal Symptoms as Assessed by the Simpson Angus Neurological Rating Scale (SAS)
Description: The best and worst possible overall scores are 40 and 0 units on a scale, respectively.
Time Frame: Baseline to 12 weeks
Population: Last Observation Carried Forward (LOCF) was used as the imputation technique.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Valproate
Number analyzed (Participants) | 15
scores on a scale | -0.6 (1.724)
Statistical Analysis 1: Comparison: Valproate; The 1 sided t-test was applied to the scores at baseline vs. the scores at 12 weeks; Test type: Superiority or Other; p = 0.199, t-test, 1 sided

9. Secondary Outcome: Tolerability as Assessed by Weight Change
Time Frame: Baseline to 12 weeks
Population: All available data was used implementing LOCF.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Valproate
Number analyzed (Participants) | 18
kilograms | 1.1 (3.6)
Statistical Analysis 1: Comparison: Valproate; The t-test was applied to the values at baseline vs. the values at 12 weeks; Test type: Superiority or Other; p = 0.21, t-test, 2 sided

10. Secondary Outcome: Tolerability as Measured by Mean Serum Level at Study Endpoint
Time Frame: Baseline to 12 weeks
Population: Last Observation Carried Forward (LOCF) was used as the imputation technique.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Valproate
Number analyzed (Participants) | 20
ug/mL | 40.86 (25.29)

ADVERSE EVENTS:
Arm/Group | Valproate
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
The findings of this study must be interpreted cautiously given the limitations of small sample size, open-label, add-on design and lack of a control or comparator group. The mean age of 61 years is not representative of the "old-old" populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes